CLINICAL TRIAL: NCT04729972
Title: Phase II, Multicenter, Open-label Safety Study of Bilateral NT-501 in Participants With Macular Telangiectasia Type 2
Brief Title: Safety Study to Evaluate Bilateral CNTF Implants in Subjects With MacTel Type 2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neurotech Pharmaceuticals (Industry)
Collaborators: The Lowy Medical Research Institute Limited (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NTMT-02B
Record Dates: First submitted 2021-01-25; First posted 2021-01-29 (Actual); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Macular Telangiectasia Type 2
Keywords: Macular Telangiectasia Type 2; CNTF; Mactel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- NT-501 in Fellow Eye (Experimental): NT-501 was implanted on Day 0 in the fellow eye of subjects who received a single NT-501 in a previous study; subjects were followed for 6 months post-implantation of NT-501 in this study.
  Interventions: Combination Product: NT-501 CNTF implant

INTERVENTIONS:
Combination Product: NT-501 CNTF implant — Single implantation of CNTF-secreting NT-501 device into fellow (untreated) eye

SUMMARY:
This is a multi-center, open-label, 6-month study to evaluate the safety of bilateral CNTF implants in participants with Macular Telangiectasia Type 2.

DETAILED DESCRIPTION:
This was a multicenter, open-label study designed to evaluate the safety of bilateral NT-501 in subjects with MacTel. All subjects who received NT-501 in a single eye prior to or in the Phase 1/2 extension study (NTMT-01/02E) or in 1 of the 2 Phase 3 studies (NTMT-03-A or NTMT-03-B), and met all other eligibility criteria, qualified for participation in the current study; enrolled subjects underwent intraocular implantation of NT-501 in the fellow eye and were followed for 6 months. Note that, throughout this report, all references to "study eye" mean the eye that received NT-501 in the current study (ie, not the eye that was treated in the previous study).

ELIGIBILITY:
General Inclusion Criteria

1. Participants from the NTMT-03 study must have completed the Month-24 visit
2. Participant in the MacTel Phase 1/2 extension (NTMT-01/02E) study or the Phase 3 study must exit these studies prior to entering the Bilateral Implant safety study (NTMT-02B)
3. Participant must be willing and able to follow the study instructions and be willing and able to complete all required study procedures and visits
4. Participant must be willing and able to provide a signed Informed Consent, as well as written documentation in accordance with the relevant country and local privacy requirements, e.g., written data protection consent
5. Females of childbearing potential must consent to a pregnancy test before entering the study
6. A participant's refusal to allow the collection of blood samples for analysis of serum CNTF, serum Ab or Nab to CNTF, Ab to NTC-201.6A cells and Ab to DFHR levels in one eye will not exclude the participant from study participation

Ocular Inclusion Criteria

1. Participant must have a positive diagnosis of MacTel type 2 with evidence of fluorescein leakage typical of MacTel and at least one of the other features that include hyperpigmentation that is outside of a 500-micron radius from the center of the fovea, retinal opacification, crystalline deposits, right-angle vessels, or inner/outer lamellar cavities in the study eye
2. Participant must have steady fixation in the foveal or parafoveal area in the study eye and sufficiently clear media for good quality photographs

General Exclusion Criteria

1. Females of childbearing potential (those who are not surgically sterilized or post- menopausal, i.e., absence of menstruation for 12 months or longer) may not participate in the study if any of the following conditions exists:

   * Pregnant (positive pregnancy test at Visit 1 or intend to become pregnant during the study)
   * Nursing (lactating)
   * Do not agree to use adequate birth control methods for the duration of the study and until 90 days after the last administration of study drug (adequate birth control methods are: hormonal - oral, implantable, transdermal or injectable contraceptives; mechanical - spermicide in conjunction with a barrier such as condom or diaphragm, intrauterine device [IUD] or surgical sterilization of partner, or total sexual abstinence)
2. Participant is too ill to likely complete the entire study, based on the investigator's assessment
3. Participant, in the opinion of the investigator, is not suitable for study participation
4. Participant with any screening laboratory finding (serum chemistry, hematology, urinalysis) that in the opinion of the investigator is not suitable for study participation
5. Participant has a history or current evidence of severe hypersensitivity to the NT-501 implant
6. Participant has a history or current evidence of a medical condition (systemic or ophthalmic disease, metabolic dysfunction, physical examination finding or clinical laboratory finding) that may in the opinion of the investigator preclude the safe administration of the NT-501 implant or adherence to the scheduled study visits, safe participation in the study or affect the results of the study (e.g., unstable or progressive cardiovascular, cerebral vascular, pulmonary, Parkinson's, liver or renal disease; depression, cancer, or dementia

Ocular Exclusion Criteria

1. Participant has a history or evidence of the following surgeries/procedures in the study eye, as assessed at Visit 1, including:

   * Submacular surgery
   * Vitrectomy
   * Retinal detachment
   * Incisional glaucoma surgery
   * Trabeculectomy or trabeculoplasty
   * Cataract surgery or laser-assisted in situ keratomileusis (LASIK) performed in the previous 6 months
2. Participant has uncontrolled glaucoma; or ocular hypertension, i.e., IOP ≥ 25 mmHg in the study eye
3. Participant has evidence of intraretinal or subretinal neovascularization or central serous chorioretinopathy in the study eye
4. Participant has evidence of ocular disorder(s) in the study eye of a severity that could confound the interpretation of study results, compromise visual acuity or require medical or surgical intervention during the study period, including retinal vascular occlusion, severe nonproliferative or proliferative diabetic retinopathy, retinal detachment, macular hole, geographic atrophy, intraretinal or subretinal neovascularization, central serous chorio-retinopathy, pathological myopia
5. Participant has a vitreous hemorrhage in the study eye at Visit 1 (Screening)
6. Participant has a spherical equivalent of the refractive error in the study eye demonstrating more than 8 diopters of myopia
7. Participant has a history or evidence of penetrating ocular trauma in the study eye
8. Participant has an anticipated need for cataract extraction in the study eye within 6 months of Visit 1 (Screening) such as cortical opacity > standard 3, posterior subcapsular opacity > standard 2, or a nuclear opacity > standard 3 as measured on the Age-Related Eye Disease Study (AREDS) clinical lens grading system
9. Participant has uveitis, history of uveitis in either eye or history of ocular herpes virus in either eye
10. Participant has undergone major surgery within the last 6 months (systemic or ocular in either eye) or who are likely to require major surgery within 6 months of Visit 1 (Screening)
11. Participant has periocular or ocular/intraocular infection or inflammation in either eye (such as infectious conjunctivitis, keratitis, scleritis, endophthalmitis) within 3 months prior to Visit 1 (Screening)
12. Participant has ocular hypotension in either eye (<6 mmHg) that in the opinion of the Investigator would interfere with the NT-501 implant insertion
13. Participant has a history of scleritis, scleral thinning, periocular, ocular, or intraocular infection or inflammation, cicatrizing conjunctival diseases any other ocular conditions in the study eye that could interfere with or complicate the surgery associated with NT-501implant insertion

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-07-21 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Aaberg, Jr, MD, Study Director — Neurotech Pharmaceuticals, LLC
Locations (10):
- United States (7):
  - Jules Stein Eye Institute, Los Angeles, California
  - National Eye Institute, Washington D.C., District of Columbia
  - Bascom Palmer, Miami, Florida
  - Massachusetts Eye and Ear Infirmary, Retina Service, Boston, Massachusetts
  - University of Michigan, Kellogg Eye Center, Ann Arbor, Michigan
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Retina Consultants of Texas, Houston, Texas
- Australia (3):
  - Save Sight Institute, Sydney, New South Wales
  - Centre for Eye Research Australia, East Melbourne, Victoria
  - Lions Eye Institute, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Chew EY, Clemons TE, Jaffe GJ, Johnson CA, Farsiu S, Lad EM, Guymer R, Rosenfeld P, Hubschman JP, Constable I, Wiley H, Singerman LJ, Gillies M, Comer G, Blodi B, Eliott D, Yan J, Bird A, Friedlander M; Macular Telangiectasia Type 2-Phase 2 CNTF Research Group. Effect of Ciliary Neurotrophic Factor on Retinal Neurodegeneration in Patients with Macular Telangiectasia Type 2: A Randomized Clinical Trial. Ophthalmology. 2019 Apr;126(4):540-549. doi: 10.1016/j.ophtha.2018.09.041. Epub 2018 Oct 4. PMID 30292541

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of the 33 enrolled subjects, 32 (97.0%) received NT-501; the exception was a subject whose surgery was canceled due to an event of arterial fibrillation that occurred prior to surgery and resulted in subject discontinuation. No subject had NT-501 removed from either eye during the study, and all 32 subjects who received NT-501 in this study completed the study.
Pre-assignment Details: Eligible subjects must have had a positive diagnosis of MacTel and previously received NT-501 in one eye prior to or in the Phase 1/2 extension study (NTMT-01/02E) or in 1 of the 2 Phase 3 studies (NTMT-03-A or NTMT-03-B). Subjects who participated in the Phase 3 study must have completed the Month 24 visit in that study and subjects enrolled in either the Phase 1/2 extension study or the Phase 3 study must have discontinued prior to enrollment in the current study.
Period: Overall Study
Arm/Group | NT-501 in Fellow Eye
Started | 33
NT-501 Implanted in Study Eye | 32
Completed | 32
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographics and characteristics are based on total number of participants who completed NT-501 implant in study eye
Arm/Group | NT-501 in Fellow Eye
Number analyzed (Participants) | 32
Age, Customized [Mean (Standard Deviation); unit: years]
  Age (Years) | 63.0 (6.55)
Age, Customized [Count of Participants; unit: Participants] — Age Groups of 50 to < 60, 60 to < 70, and greater than or equal to 70
  Participants
    50 to < 60 years | 9
    60 to < 70 years | 17
    > or = to 70 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 0
  Unknown or Not Reported | 1
BCVA (letters) for Study Eye [Mean (Standard Deviation); unit: letters correctly read] — Baseline letter score using the standard Treatment Diabetic Retinopathy Study (ETDRS) chart
  letters correctly read
    Study Eye | 68.7 (11.01)
    Fellow Eye | 70.1 (9.58)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Ocular and/or Non-ocular Treatment Emergent Adverse Events
Description: Assess the incidence and severity of adverse events (AEs) following bilateral ocular implantation of NT-501
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | NT-501 in Fellow Eye
Number analyzed (Participants) | 32
Participants
  At least 1 TEAE | 26
  At least 1 ocular TEAE in study eye | 26
  At least 1 ocular TEAE in fellow eye | 6
  At least 1 nonocular TEAE | 13
  At least 1 treatment related ocular TEAE | 26
  At least 1 treatment related nonocular TEAE | 0
  At least 1 SAE | 2
  NT-501 removal from either eye | 0

2. Secondary Outcome: Serum Levels of CNTF and Immunogenicity for NT-501
Description: Incidence of positive serum levels of CNTF and immunogenicity for NT-501 with quantification of antibodies (Ab) to CNTF, neutralizing antibodies (NAb) to CNTF, Ab to NTC-201-6A cells, and Ab to mouse dihydrofolate reductase (mDHFR) at any time.
Time Frame: 6 months
Population: A neutralizing antibody test to NT-501-produced CNTF was performed to verify or refute CNTF antibody detected in one participant. The neutralizing antibody test refuted that the antibody detected was to NT-501 CNTF.
Measure: Count of Participants; unit: Participants
Arm/Group | NT-501 in Fellow Eye
Number analyzed (Participants) | 32
Participants
  CNTF Positive | 0
  Ab Positive to CNTF | 1
  Neutralizing Ab to CNTF | 0
  Ab to NTC | 0
  ab to DHRF | 0

ADVERSE EVENTS:
Time Frame: Through 6 months post implant
Arm/Group | NT-501 in Fellow Eye
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 2/32
Other Adverse Events (participants affected / at risk) | 26/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-501 in Fellow Eye (N=32)
Device Extrusion (Surgical and medical procedures) | 1 (1)
Feces discolored (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-501 in Fellow Eye (N=32)
Eye pain (Eye disorders) | 9 (9)
Ocular discomfort (Eye disorders) | 9 (9)
Conjunctival haemorrhage (Eye disorders) | 8 (8)
Eye irritation (Eye disorders) | 4 (4)
Dry eye (Eye disorders) | 2 (2)
Anterior chamber cell (Eye disorders) | 1 (1)
Anterior chamber flare (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Cataract subcapsular (Eye disorders) | 1 (1)
Conjunctival hyperaemia (Eye disorders) | 1 (1)
Conjunctival oedema (Eye disorders) | 1 (1)
Conjunctivitis allergic (Eye disorders) | 1 (1)
Corneal pigmentation (Eye disorders) | 1 (1)
Delayed dark adaptation (Eye disorders) | 1 (1)
Epiretinal membrane (Eye disorders) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1)
Foreign body sensation in eyes (Eye disorders) | 1 (1)
Halo vision (Eye disorders) | 1 (1)
Iris transillumination defect (Eye disorders) | 1 (1)
Iritis (Eye disorders) | 1 (1)
Photophobia (Eye disorders) | 1 (1)
Photopsia (Eye disorders) | 1 (1)
Punctate keratitis (Eye disorders) | 1 (1)
Retinal haemorrhage (Eye disorders) | 1 (1)
Vitreous detachment (Eye disorders) | 1 (1)
Vitreous haemorrhage (Eye disorders) | 1 (1)
Allergy to sutures (Immune system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 1 (1)
Intraocular pressure decreased (Investigations) | 1 (1)
Pyogenic granuloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Device extrusion (Product Issues) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-01-21): https://cdn.clinicaltrials.gov/large-docs/72/NCT04729972/Prot_001.pdf
  • Statistical Analysis Plan (2022-07-14): https://cdn.clinicaltrials.gov/large-docs/72/NCT04729972/SAP_002.pdf